CLINICAL TRIAL: NCT00328029
Title: Assessment of Respiratory Functions After a Conditioning Regimen With Busulfan for Allograft or Autograft in a Unicenter Pediatric and Prospective Population
Brief Title: Respiratory Side Effects of Busulfan High Dose Chemotherapy in a Pediatric Population
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER, Direction de la Recherche Clinique et de l'Innovation - Hôpitaux Universitaires de Strasbourg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2999
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Signs and Symptoms, Respiratory
Keywords: Busulfan; pharmacokinetic; respiratory function assessment; Busulfan pharmacokinetic and respiratory function tests
MeSH Terms: conditions — Signs and Symptoms, Respiratory | interventions — Busulfan; Respiratory Physiological Phenomena; Transplantation, Autologous; Pharmacokinetics

INTERVENTIONS:
Drug: busulfan — 5mg/kg/day (oral route : 4 doses/day for 4 days)
Procedure: respiratory function tests — respiratory function tests before allograft or autograft and at several times in the follow up (3, 6, 12, 18 and 24 months).
  Other Names: before allograft or autograft and at several times in the follow up (3, 6, 12, 18 and 24 months).
Procedure: pharmacokinetics, done during the treatment — 12 blood collections :
  * after 1st Busulfan taken : t0; t0 + 30 mn; t0 + 1h; t0 + 2h ; t0 + 3h ; t0 + 4h ; t0 + 5 h.
  * 3 hours after 2nd taken of Busulfan
  * 3 hours after 3rd taken of Busulfan
  * 3 hours after 4th taken of Busulfan
  * 3 hours after 5th taken of Busulfan
  * 3 hours after 6th taken of Busulfan.

SUMMARY:
Recently, several conditioning regimens did not include total body irradiation (TBI) anymore, especially in the case of young children due to cognitive sequelae and late effects on growth and height. Thus, such effective chemotherapy conditioning regimens were developed to avoid these complications. Busulfan is one of the major drugs used in these treatments, but, is also administered in high dose chemotherapy followed by autograft. In both situations, long term pulmonary side effects were diagnosed in a few cases. Even if the occurrence is not very frequent, the clinical management is a real challenge regarding the reduced quality of life and life expectancy of these patients. Up to now, no correlation was done between respiratory sequelae and busulfan pharmacokinetics. Hence, in the investigators' pediatric onco-hematological unit, a prospective study will begin and last three years to assess the respiratory side effects due to busulfan and their potential links with individual drug pharmacokinetic measures. These results will be compared to patients treated with TBI during the same period of time.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 3 years old treated by busulfan or TBI in their conditioning regimens before allograft or busulfan in high dose chemotherapeutic regimens followed by autograft will be included after parents informed assent.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2006-07; Primary Completion 2012-01 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Determination of respiratory side effect frequency in the two years follow up of allograft or autograft treated with busulfan | before allograft or autograft and at several times in the follow up (3, 6, 12, 18 and 24 months).

SECONDARY OUTCOMES:
Comparison to respiratory side effect frequency with TBI conditioning regimen | before allograft or autograft and at several times in the follow up (3, 6, 12, 18 and 24 months).
Busulfan pharmacokinetics | after 1st Busulfan taken : t0; t0 + 30 mn; t0 + 1h; t0 + 2h ; t0 + 3h ; t0 + 4h ; t0 + 5 h ; 3 h after 2nd Busulfan taken ; 3 hours after 3rd Busulfan taken ; 3 h after 4st Busulfan taken ;3 h after 5st Busulfan taken ;3 h after 6st Busulfan taken
Establish a potential link between respiratory side effects and busulfan pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Lutz, MD, Study Director — Service de Pédiatrie Onco-Hématologie - Hôpital de Hautepierre
Locations (2):
- France (2):
  - Service d'Explorations Fonctionelles Respiratoires - Hôpital Civil, Strasbourg
  - Service de Pédiatrie Onco-Hématologie - Hôpital de Hautepierre, Strasbourg